CLINICAL TRIAL: NCT01416974
Title: A Phase I Trial of Consolidation Therapy With Autologous T Cells Genetically Targeted to the B Cell Specific Antigen CD19 in Patients With Chronic Lymphocytic Leukemia Following Upfront Chemotherapy With Pentostatin, Cyclophosphamide and Rituximab
Brief Title: Consolidation Therapy With Autologous T Cells Genetically Targeted to the B Cell Specific Antigen CD19 in Patients With Chronic Lymphocytic Leukemia Following Upfront Chemotherapy With Pentostatin, Cyclophosphamide and Rituximab
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-048
Record Dates: First submitted 2011-08-12; First posted 2011-08-15 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Leukemia
Keywords: 19-28Z RETROVIRUS; CYCLOPHOSPHAMIDE (CYTOXAN); autologous T cells; Leukapheresis; 11-048
MeSH Terms: conditions — Leukemia | interventions — Cyclophosphamide

ARMS (1):
- consolidative therapy with autologous T cells genetically (Experimental): A phase I trial of consolidation therapy with autologous T cells genetically targeted to the B cell specific antigen CD19 for patients with chronic lymphocytic leukemia following upfront chemotherapy with pentostatin, cyclophosphamide and rituximab.
  Interventions: Drug: cyclophosphamide; Biological: modified T cells

INTERVENTIONS:
Drug: cyclophosphamide — Patients will first receive a single infusion of therapy conditioning with cyclophosphamide.
Biological: modified T cells — followed by consolidative therapy with the modified T cells in 3 planned cohorts.

SUMMARY:
The purpose of this Phase I study is to test the safety and effect of specially prepared cells collected from the patients called "modified T cells." We want to find a safe dose of modified T cells for patients who have disease remaining after initial chemotherapy. We also want to find out what effects these T cells have on you and your leukemia.

ELIGIBILITY:
Inclusion Criteria:

* CLL patients with evidence of residual disease, who have achieved PR, nPR or CR with detectable MRD following upfront therapy consisting of pentostatin, cyclophosphamide and rituximab.
* The presence of MRD will be assessed by the flow cytometry and polymerasechain reaction at the MSKCC Diagnostic Molecular Pathology Laboratory.
* Age ≥ 18 years of age.
* Creatinine ≤2.0 mg/100 ml, bilirubin ≤2.0 mg/100 ml, AST and ALT ≤3.0x normal, PT and PTT ≤2x normal outside the setting of stable chronic anticoagulation therapy, absolute neutrophil count ≥500/mm3, platelets ≥50,000/mm3, hemoglobin ≥8.0g/dl with transfusion support.
* Adequate pulmonary function as assessed by ≥92% oxygen saturation on room air by pulse oximetry.

Exclusion Criteria:

* Karnofsky performance status <70.
* Pregnant or lactating women. Women and men of childbearing age should use effective contraception while on this study and continue for 1 year after all treatment is finished.
* Impaired cardiac function (LVEF <40%) as assessed by ECHO or MUGA scan.
* Patients previously treated with allogeneic bone marrow or stem cell transplantation are ineligible.
* Patients who are immediate candidates for allogeneic bone marrow or stem cell transplantation. Patients who refuse this option remain eligible and need to be documented as such in patient medical record.
* CLL patients with transformed disease (Richter's transformation) are ineligible for enrollment on this study.
* Patients with following cardiac conditions will be excluded:
* New York Heart Association (NYHA) stage III or IV congestive heart failure
* Myocardial infarction ≤6 months prior to enrollment
* History of clinically significant ventricular arrhythmia or unexplained syncope, not believed to be vasovagal in nature or due to dehydration
* History of severe non-ischemic cardiomyopathy with EF ≤20%
* Patients with HIV and active hepatitis B or hepatitis C infection are ineligible.
* Patients with any concurrent active malignancies as defined by malignancies requiring any therapy other than expectant observation, with the exception of squamous and basal cell carcinoma of skin.

STEP 2 REGISTRATION (Treatment):

The following additional criteria must be met in order for a patient to be eligible to receive the modified T cell infusion. These labs are to be obtained within 2 weeks of T cell infusion.

* Creatinine ≤2.0 mg/100 ml, bilirubin ≤2.0 mg/100 ml, AST and ALT ≤3.0x normal, PT and PTT ≤2x normal outside the setting of stable chronic anticoagulation therapy, absolute neutrophil count ≥500/mm3, platelets ≥50,000/mm3, hemoglobin ≥8.0g/dl with transfusion support.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-08-22 (Actual); Primary Completion 2019-01-07 (Actual); Study Completion 2019-01-07 (Actual)

PRIMARY OUTCOMES:
toxicity | 2 years
  Criteria for toxicity: Toxicity will be graded on a scale of 1 to 5 as described by the NCI Common Terminology Criteria for Adverse Events (CTCAE), version 3.0
maximum tolerated dose (MTD) | 2 years
  If none of the initial 3 patients in a cohort experience a dose limiting toxicity (DLT) then the next dose level will be studied in another cohort of 3 patients

SECONDARY OUTCOMES:
disease response | 2 years
  The major criteria for determination of response to therapy in patients with CLL include physical examination and examination of the peripheral blood and bone marrow. Radiographic studies are not required but those that were abnormal pre-treatment will be repeated to document the degree of maximal response.
change in cellular and cytokine tumor microenvironment | 2 years
  Cellular tumor microenvironment analysis: The presence of regulatory T cells (Tregs) and myeloid derived suppressor cells (MDSCs), as well as the presence of immune effector cells including dendritic cells, NK cells, and effector T cells will be assessed by fluorescence-activated cell sorting (FACS).
the impact of infused modified T cells | 2 years
  Persistence of gene-modified T cells is defined by the presence of any percentage of detectable cells. The percentage of gene-modified T cells/ total T cells will be recorded for all patients treated at each dose level. In addition, gene-modified T cells will be measured daily for two days, weekly for eight weeks and monthly for six months (by FACS and RT-PCR).

CONTACTS AND LOCATIONS:
Overall Officials: Jae Park, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm